CLINICAL TRIAL: NCT04953338
Title: The Mental Health Associations With Vitiligo: a Population-based Cohort Study in the UK
Brief Title: Mental Health Associations With Vitiligo
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: P044
Record Dates: First submitted 2021-06-19; First posted 2021-07-07 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Vitiligo; Depressive Episode; Recurrent Depressive Disorder; Anxiety Disorders; Social Phobia; Adjustment Disorders; Substance Abuse; Self-Harm, Deliberate; Overdose; Suicide, Attempted; Parasuicide
MeSH Terms: conditions — Vitiligo; Depressive Disorder; Anxiety Disorders; Phobia, Social; Adjustment Disorders; Substance-Related Disorders; Self-Injurious Behavior; Drug Overdose; Suicide, Attempted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with a confirmed diagnosis of Vitiligo within the study period will be included as cases for analysis.
  Interventions: Other: Exposure of mental health condtion of interest
- Controls: The controls will be defined by matching cases with people who have never been diagnosed with vitiligo either prior to or during the study period, by age and sex, at General Practice level.
  Interventions: Other: Exposure of mental health condtion of interest

INTERVENTIONS:
Other: Exposure of mental health condtion of interest — Common mental health conditions consist of depressive episodes, recurrent depressive disorder and anxiety disorder.

SUMMARY:
This cohort study is a large population-based study in the UK to determine the risks of comorbid mental health conditions (including depression, anxiety and other potential psychological complications of vitiligo) in adults with vitiligo compared to controls and to evaluate whether the relative risks may vary by different ethnicity.

DETAILED DESCRIPTION:
This study has two primary outcomes 1) Prevalence and incidence of mental health condtions in people diagnosed with vitiligo compared to matched controls and 2) Primary care and secondary healthcare utilisation in patients diagnosed with vitiligo and having a prevalent depressive conditon compared to matched controls. In addition, the study examines risk of time off work and unemployment in people diagnosed with vitiligo compared to matched controls.

ELIGIBILITY:
Inclusion Criteria:

* All eligible adults ≥18 (as at date of vitiligo diagnosis for cases or start of follow-up for controls) registered with GP practices contributing data to OPCRD between January 1, 2004 and December 31, 2020, were eligible for inclusion in the study.

Exclusion Criteria:

* People with less than 1 year of follow up available

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will use routinely collected and collated data from OPCRD to provide a broadly representative sample of the population of the UK.
Sampling Method: Non-Probability Sample
Enrollment: 36104 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data Ltd
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
OPCRD data can be accessed by bone fide researchers for specific research projects subject to approval by Anonymised Data Ethics & Protocol Transparency (ADEPT) Committee. The data utilised for this study cannot be made available without such approval.
Supporting Information: Study Protocol
Time Frame: The data will be available subject to approvals for two years after the study publication date
Access Criteria: Data sharing is subject to ADEPT committee approval

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases | Controls
Started | 7224 | 28880
Completed | 7224 | 28880
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 7224 | 28880 | 36104
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [33 to 58] | 44 [32 to 58] | 44 [32 to 58]
Age, Customized [Count of Participants; unit: Participants]
  Age group, years: 18-29 | 1377 | 5534 | 6911
  Age group, years: 30-39 | 1526 | 6087 | 7613
  Age group, years: 40-49 | 1463 | 5822 | 7285
  Age group, years: 50-59 | 1251 | 5006 | 6257
  Age group, years: 60-69 | 918 | 3647 | 4565
  Age group, years: 70-76 | 534 | 2155 | 2689
  Age group, years: 80+ | 155 | 629 | 784
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3828 | 15304 | 19132
  Male | 3396 | 13576 | 16972
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3504 | 14013 | 17517
  Asian or Asian British | 1060 | 3200 | 4260
  Black, African, Caribbean or Black British | 170 | 556 | 726
  Mixed | 66 | 238 | 304
  Other | 259 | 1155 | 1414
  Not stated | 199 | 949 | 1148
  Missing | 1966 | 8769 | 10735
Body Mass Index, Categorical [Count of Participants; unit: Participants] — Body Mass Index (BMI) is a based on a participants height and weight.
  Participants
    <18.5 Underweight | 174 | 670 | 844
    18.5-24.9 Healthy weight | 2129 | 7544 | 9673
    25-29.9 Overweight | 2282 | 8511 | 10793
    30-34.9 Class I obesity | 1080 | 4316 | 5396
    35-39.9 Class II obesity | 367 | 1674 | 2041
    >40 Class III obesity | 211 | 1013 | 1224
    Not recorded | 981 | 5152 | 6133
Smoking Status, Categorical [Count of Participants; unit: Participants]
  Non-smoker | 2357 | 8629 | 10986
  Current smoker | 1147 | 5881 | 7028
  Ex-smoker | 3521 | 12862 | 16383
  Passive smoker | 30 | 77 | 107
  Not recorded | 169 | 1431 | 1600
Alcohol use, Categorical [Count of Participants; unit: Participants]
  Non-drinker | 2438 | 8984 | 11422
  Safe use | 2799 | 11101 | 13900
  Excess use | 970 | 3604 | 4574
  Alcoholism | 116 | 499 | 615
  Not recorded | 901 | 4692 | 5593

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Depressive Episodes
Description: Prevalence of common mental health conditions (depressive episodes) in adult people diagnosed with vitiligo and matched controls without vitiligo.
Time Frame: At the time of diagnosis in all people diagnosed with vitiligo 2004-2020 inclusive. For matched controls, the date of diagnosis of their matched case.
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 7224 | 28880
Participants | 1018 | 4007

2. Primary Outcome: Risk of Depressive Episodes Within Adult Patients With Vitiligo
Description: Adjusted hazard ratio calculated using Cox proportional hazards models
Time Frame: Within two years of vitiligo diagnosis. For matched controls, within two years of the date of diagnosis of their matched case.
Population: Patients with a pre-existing diagnosis of depressive episodes were excluded from this analysis
Measure: Count of Participants; unit: Participants
Groups:
- Controls (reference group): The controls will be defined by matching cases with people who have never been diagnosed with vitiligo either prior to or during the study period, by age and sex, at General Practice level.
Arm/Group | Cases | Controls (reference group)
Number analyzed (Participants) | 6206 | 21602
Participants | 157 | 501
Statistical Analysis 1: Comparison: Controls (reference group); Test type: Superiority; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.92 to 1.32] — Calculated as the relative risk of a person diagnosed with vitiligo having a depression episode versus people not diagnosed with vitiligo

3. Primary Outcome: Number of Participants With Anxiety Disorder
Description: Prevalence of common mental health conditions (Anxiety Disorder) in adult people diagnosed with vitiligo and matched controls without vitiligo.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 7224 | 28880
Participants | 569 | 2031

4. Primary Outcome: Number of Participants With Recurrent Depressive Disorder
Description: Prevalence of common mental health conditions (Recurrent Depressive Disorder) in adult people diagnosed with vitiligo and matched controls without vitiligo.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 7224 | 28880
Participants | 1093 | 4305

5. Primary Outcome: Risk of Anxiety Disorder Within Adult Patients With Vitiligo
Description: Adjusted hazard ratio calclulated using Cox Proportional hazard models
Time Frame: as for outcome 2
Population: Patients with a pre-existing diagnosis of anxiety disorder were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls (reference group)
Number analyzed (Participants) | 6655 | 24834
Participants | 122 | 382
Statistical Analysis 1: Comparison: Controls (reference group); Test type: Superiority; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [1.01 to 1.51] — Calculated as the relative risk of a person diagnosed with vitiligo having with anxiety disorder versus people not diagnosed with vitiligo

6. Primary Outcome: Risk of Recurrent Depressive Disorder Within Adult Patients With Vitilgo
Description: Adjusted hazard ratio calculated using Cox proportional hazards models. Adjusted for age, gender, ethnicity, social deprivation quintile, body mass index, smoking status, alcohol use and comorbidities (hypertension, hyperlipidaemia, type 2 diabetes, atrial fibrillation, angina, myocardial infarction, heart failure, stroke, chronic kidney disease stages 3-5, chronic obstructive pulmonary disease, asthma, chronic liver disease and dementia).
Time Frame: as for outcome 2
Population: Patients with a pre-existing diagnosis of recurrent depressive disorder were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls (reference group)
Number analyzed (Participants) | 6131 | 21091
Participants | 113 | 312
Statistical Analysis 1: Comparison: Controls (reference group); Test type: Superiority; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [1.01 to 1.56] — Calculated as the relative risk of a person diagnosed with vitiligo having with recurrent depressive disorder versus people not diagnosed with vitiligo

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and nonserious adverse events were not assessed for study participant.
Arm/Group | Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT04953338/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT04953338/SAP_001.pdf